CLINICAL TRIAL: NCT05566600
Title: Epicardial Injection of Allogeneic Human Pluripotent Stem Cell-derived Cardiomyocytes to Treat Severe Chronic Heart Failure
Brief Title: Allogeneic iPSC-derived Cardiomyocyte Therapy in Patients With Worsening Ischemic Heart Failure
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Help Therapeutics (Industry)
Collaborators: Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JFYang
Record Dates: First submitted 2022-09-22; First posted 2022-10-04 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Ischemic Heart Failure; Chronic Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dose level 1 (Experimental): 100 million iPSC-CMs administration
  Interventions: Biological: Human (allogeneic) iPS-cell-derived cardiomyocyte
- Dose level 2 (Experimental): 200 million iPSC-CMs administration
  Interventions: Biological: Human (allogeneic) iPS-cell-derived cardiomyocyte
- Dose level 3 (Experimental): 400 million iPSC-CMs administration
  Interventions: Biological: Human (allogeneic) iPS-cell-derived cardiomyocyte
- Control (No Intervention): Participants will received CABG surgery only

INTERVENTIONS:
Biological: Human (allogeneic) iPS-cell-derived cardiomyocyte — 10-20 epicardial injections (0.25 mL each) of iPSC-CMs will be delivered in the border zone of the infarcted myocardium
  Arms: Dose level 1; Dose level 2; Dose level 3

SUMMARY:
This study is designed to evaluate the safety and efficacy of allogeneic induced pluripotent cell derived cardiomyocytes (iPSC-CMs) in treating patients with worsening ischemic heart failure undergoing coronary artery bypass graft surgery.

After screening, iPSC-CMs will be administrated intramyocardially in consented and eligible patients undergoing open-chest CABG surgery and the estimated population size for the study will be 32 patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged 35-75 (including 35 and 75).
* Signed the Informed Consent Form (ICF).
* Have chronic left ventricular dysfunction.
* Have NYHA Class III-IV cardiac function even after improved medication for the treatment of advanced chronic heart failure.
* Have indications for Coronary Artery Bypass Grafting.
* LVEF < 40% as determined by echocardiogram (data collected up to 6 months prior to inclusion evaluation are valid; data collected within 1 month since a myocardial infarction are invalid).
* Weakening or absence of segmental regional wall motion as determined by standard imaging

Exclusion Criteria:

* PRA ≥ 20% or DSA-positive
* Patient received ICD transplantation, CRT or similar treatment.
* Patients with valvular heart disease or received heart valvular disease
* Patients received treatment of percutaneous transluminal coronary intervention (PCI)
* Patients with atrial fibrillation
* Patients previously suffered sustained ventricular tachycardia or sudden cardiac death.
* Baseline glomerular filtration rate <30ml/min/1.73m2.
* Liver dysfunction, as evidenced by enzymes (AST and ALT) greater than three times the ULN.
* Hematological abnormality: A hematocrit <25% as determined by HCT, white blood cell<2500/ul or platelet values <100000/ul without another explanation.
* Known, serious radiographic contrast allergy, penicillin allergy, streptomycin allergy.
* Coagulopathy (INR>1.3) not due to a reversible cause.
* Contra-indication to performance of a MRI scan.
* Recipients of organ transplant.
* Clinical history of malignancy within 5 years (patients with prior malignancy must be disease free for 5 years).
* Non-cardiac condition that limits lifespan <1 year.
* On chronic therapy with immunosuppressant medication, such as glucocorticoid and TNFα antagonist.
* Patients allergy to or cannot use immunosuppressant.
* Serum positive for HIV, HBV, HCV, TP.
* Currently enrolled other investigational therapeutic or device study.
* Patients who are pregnant or breast feeding.
* Other conditions that researchers consider not suitable to participate in this study.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-10-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety in terms of the incidence and severity of adverse events | within 1 month post CABG surgery
  Number of participants with death, fatal myocardial infarction, stroke, ventricular tachycardia sustained for >15 seconds and newly formed tumor

SECONDARY OUTCOMES:
Incidence of adverse events | 1~6 months post CABG surgery
  Adverse events that require medical intervention
Cardiac assessment | 1~6 months post CABG surgery
  24-hour Holter Monitoring post the CABG surgery
Incidence of newly formed tumor | 1~12 months post CABG surgery
  Evaluation by chest, abdominal and pelvic CT scan and PET-CT scan
Immunogenic assessments | 1 month, 3 months and 6 months post CABG surgery
  Donor specific antibody (DSA), serum anti-human leukocyte antigens (anti-HLA) antibody/panel-reactive antibody (PRA) serology monitoring
Changes in left ventricle function evaluation by echocardiogram (ECHO) or cardiac MRI | from baseline to 12 months at 3, 6, and 12 months post CABG surgery
  Changes in cardiac function will be assessed by left ventricular end-systolic volume (LVESV, mL) changes from baseline to 12 months post surgery
Changes in 6-minute walk test (6MWT) | from baseline to 12 months at 1, 3, 6, and 12 months post CABG surgery
Changes in NYHA functional classification | from baseline to 12 months at 1, 3, 6, and 12 months post CABG surgery
Changes in quality of life (QoL) | from baseline to 12 months at 1, 3, 6, and 12 months post CABG surgery
  Quality of life changes as measured by Minnesota Living with Heart Failure Questionnaire (MLHFQ) scores
Incidence of hospitalization for worsening heart failure | 1~12 months post CABG surgery

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The second xiangya hospital of central south university, Changsha, Hunan
  - HelpThera, Nanjing, Jiangsu